CLINICAL TRIAL: NCT04541719
Title: Patient Controlled Remifentanil Analgesia vs. Epidural Analgesia for Normal Labour. A Prospective Randomised Study
Brief Title: Patient Controlled Remifentanil Analgesia for Normal Labour
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Mansoura University (Other)
Collaborators: Cairo University (Other); Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed R El Tahan, Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MFM-XYZ-2017
Record Dates: First submitted 2020-09-02; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Labor Pain; Full Term Pregnancy
MeSH Terms: conditions — Labor Pain | interventions — Analgesia, Epidural

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient-controlled remifentanil analgesia (Active Comparator): Patients will received Patient-controlled remifentanil analgesia starting from labour pain until delivery
  Interventions: Drug: Patient-controlled remifentanil analgesia
- Epidural analgesia (Placebo Comparator): Patients will received continuous epidural analgesia starting from labour pain until delivery
  Interventions: Drug: Epidural analgesia

INTERVENTIONS:
Drug: Patient-controlled remifentanil analgesia — Patient controlled remifentanil analgesia with a regimen to provide a bolus of 40 μg remifentanil with a lockout interval of 2 min
  Arms: Patient-controlled remifentanil analgesia
Drug: Epidural analgesia — Patients will receive continuous epidural analgesia using bupivacaine 0.125% in conjunction with fentanyl 2 ug/ml at a rate of 8-15 ml/hr
  Arms: Epidural analgesia

SUMMARY:
Patient controlled remifentanil analgesia might offer comparative overall patient satisfaction and improved quality of analgesia after normal labour with continuous epidural analgesia.

DETAILED DESCRIPTION:
We are aiming to study the effects of patient controlled remifentanil analgesia and epidural analgesia for normal labour in full term parturients on:

* Peripartum analgesia
* Overall patient's satisfaction
* Maternal adverse effects
* Neonatal outcomes

ELIGIBILITY:
Inclusion Criteria:

* Gestational age > 36 weeks
* American Society of Anesthesiologists physical class I to III

Exclusion Criteria:

* Allergy to study solution
* Contraindications to epidural analgesia
* Non consented parturients
* Communications barriers.
* Intrauterine foetal growth retardation
* Foetal distress

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Overall patient's satisfaction | For 24 hours after labour
  As being assesses using 100-mm visual analog score (0: unsatisfied, 100: very satisfied)

SECONDARY OUTCOMES:
Pain Visual Analog Score at rest | For 24 hours after the start of labour pain
  As being assesses using 10-cm visual analog score (0: no pain, 10: very agonising pain)
Pain Visual Analog Score on movement | For 24 hours after the start of labour pain
  As being assesses using 10-cm visual analog score (0: no pain, 10: very agonising pain)
Maternal nausea and vomiting | For 24 hours after the start of labour pain
  (0: no nausea or vomiting, 1: severe nausea, 3: vomiting)
Maternal respiratory depression | For 24 hours after the start of labour pain
  If respiratory rate decreases less than 10/min
Neonatal Apgar score at 1 min | For 5 min after birth
  Assessed using 5-points Apgar score
Neonatal Apgar score at 5 min | For 5 min after birth
  Assessed using 5-points Apgar score
Neonatal blood PaO2 | For 5 min after birth
  PaO2 value
Neonatal blood PaCO2 | For 5 min after birth
  PaCO2 value
Neonatal blood pH | For 5 min after birth
  pH value

CONTACTS AND LOCATIONS:
Overall Officials: Nabil A Abd El Raouf, MD, Study Chair — Professor in Cardiothoracic Ananesthesia
Locations (1):
- Mansoura University Hospitals, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided